CLINICAL TRIAL: NCT07169526
Title: Gesundheitskompetenz Und Selbstwirksamkeitserwartung Bei PatientInnen Mit Alkoholbedingter Leberzirrhose
Brief Title: Health Literacy and Self-efficacy Expectations in Patients With Alcohol-related Liver Cirrhosis
Acronym: GESA
Status: Recruiting | Type: Observational
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 12014-BO-K-2025; 12014-BO-K-2025 (Other: Ethikkomission Medizinsiche Hochschule Hannover)
Record Dates: First submitted 2025-09-03; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Self-Efficacy; Health Literacy; Liver Cirrhosis; ALD - Alcoholic Liver Disease
MeSH Terms: conditions — Liver Cirrhosis; Liver Diseases, Alcoholic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to quantify the health literacy and self-efficacy in people with alcohol-related liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* age (18-99)
* liver cirrhosis

Exclusion Criteria:

* pregnancy
* insufficient german

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: people with liver cirrhosis
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Level of self-efficacy at baseline, assessed using the Scale for General Self-Efficacy (Skala zur Allgemeinen Selbstwirksamkeitserwartung) | baseline
Level of health literacy at baseline, assessed using the European Health Literacy Survey Questionnaire (HLS-EU-Q47) | baseline

SECONDARY OUTCOMES:
Occurrence of hepatic decompensation or liver-related death | until end of study
Rehospitalization due to liver-related complications | Throughout study completion (up to 12 months)
Hepatic decompensation episodes | Throughout study completion (up to 12 months)
Level of quality of life, assessed using the [e.g., SF-36 Questionnaire] | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Medizinische Hochschule Hannover, Hanover, Germany